CLINICAL TRIAL: NCT06416969
Title: Stimulation of Regional Lipolysis and Adipocyte Lipolysis Proteins
Brief Title: Regional Lipolysis and Adipocyte Lipolysis Protein Stimulation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael D. Jensen, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-004069; R01DK040484 (NIH)
Record Dates: First submitted 2024-05-01; First posted 2024-05-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Somatostatin; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obesity Group (Experimental): Subjects that have upper body obesity will receive somatostatin plus epinephrine
  Interventions: Drug: Somatostatin; Drug: Epinephrine
- Lean Group (Experimental): Subject wo are normal weight will receive somatostatin plus epinephrine
  Interventions: Drug: Somatostatin; Drug: Epinephrine

INTERVENTIONS:
Drug: Somatostatin — Intravenous infusion 200 ug/hr for 2 hours, 100 ug/hr for 30 minutes
Drug: Epinephrine — Intravenous infusion

SUMMARY:
Adults who gain most of their excess weight in the abdominal area typically do not respond to factors that "turn on" fat cells the same way as people who don't have excessive weight. Researchers are trying to understand why fat tissue responds differently in people with different body types.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age who are able to comprehend instructions, follow study procedures, willing to sign an informed consent form, and consume an isoenergetic diet eating all meals from Mayo Clinical Research and Trials Unit for at least 3 days prior to study.
* Overweight/Obese volunteers will have a BMI 29.0 - 40.0 kg/m2

  o Upper body/visceral obesity (UBO) in women will be defined as those with a waist-hip ratio (WHR) > 0.85 and/or increased visceral fat by single slice CT scan, usually with > 120 cm2 of visceral fat by CT scanning or a visceral fat/total fat ratio of > 0.30, and/or biochemical evidence of metabolic syndrome as defined by adenosine triphosphate (ATP) III criteria (fasting plasma triglycerides ≥ 150 mg/dL, HDL-cholesterol < 50 mg/dL for women and < 40 mg/dL for men, fasting plasma glucose ≥ 100 mg/dL). Upper body obesity in men will be defined as a waist-hip ratio of >0.95 and/or increased visceral fat (visceral fat area > 120 cm2 or a visceral/total fat abdominal ratio by CT of > 0.40) by single slice CT scan and/or biochemical evidence of metabolic syndrome as defined by ATP III criterial. These visceral fat values are based upon the data collected at Mayo Clinic using our methods, and are correlated with dyslipidemia and hyperinsulinemia.
* Female subjects are eligible if they meet the following criteria:

  * Are not pregnant or nursing
  * All women of childbearing potential will have a negative urine pregnancy test at screening and a negative urine pregnancy test within 48 hours before administering study drug.
* Recent or current research participation in a study that involves an investigational drug. Participants in other clinical trials that involve an investigational drug will not be able to participate in this study until 12 weeks after their participation in the other study is complete or > than five half-lives of the compound, whichever is longer. If Yes look at consent form and f/u visits:
* Current use of medications that alter fatty acid or adipose metabolism possibly given: if yes, exclude
* Amount of blood drawn during the study (if our study plus this one draw ≥ 450 ml these should be separated by 8 weeks
* Previous labs:
* Fasting glucose < 126 mg/dl for non-diabetic UBO
* Hb ≥ 11.0 for women and ≥ 12 for men
* platelets > 100 000

Exclusion Criteria:

* Individuals with a history of a disease process such as:

  * Ischemic heart disease
  * Atherosclerotic valvular disease
  * Persistent blood pressure greater than 160/95 despite antihypertensive medication
  * Peripheral artery disease
  * Any history of trans-ischemic attacks.
  * Coronary artery disease.
  * Liver cirrhosis
  * Significant renal impairment as documented in medical chart.
* Smokers
* Diagnosis of Diabetes Mellitus.
* Concomitant use of medications that can alter free fatty acid metabolism or pose a drug-drug interaction: statins (if yes hold for 4 weeks and receive primary care provider's approval); Niacin; Fibrates; thiazolidinedione; Beta-blockers; Oral or injected corticosteroids or anabolic steroids; Linezolid; Dihydroergotamine; Phenelzine; daily phosphodiesterase inhibitors
* Allergy to lidocaine
* Allergy to indocyanine green.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Free Fatty Acid (FFA) release from femoral, splanchnic and upper body subcutaneous adipose tissue | approximately 3.5 hours
  regional palmitate release rates (micromol/min) will be measured using a combination of leg and splanchnic blood flow combined with stable isotope tracer measurements of palmitate uptake and release across the leg and splanchnic bed. Upper body, non-splanchnic palmitate release will be calculated as: total palmitate release - (splanchnic palmitate release + (leg palmitate release x 2)). Release rates will be measured at baseline (overnight fasting) and in response to the infusion of somatostatin plus epinephrine. This will allow us to understand the factors that may limit maximum lipolysis stimulation in upper body obesity for leg, splanchnic and upper body non-splanchnic adipose tissue palmitate release.
stimulated FFA release in volunteers with and without obesity. | approximately 3.5 hours
  we will measure whether stimulated adipose tissue lipolysis from infusions of somatostatin and epinephrine is impaired in UBO and, if so, if this is related to regional differences in lipolysis and lipolysis-regulating proteins;

SECONDARY OUTCOMES:
Role of reesterification in adipose tissue FFA release | approximately 3.5 hours
  We will measure the regional FFA:glycerol release ratio, a measure of intracellular reesterification, differs between UBO and non-UBO adults in a way that accounts for the differences in systemic FFA delivery. This will require the use of both FFA and glycerol tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jensen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No